CLINICAL TRIAL: NCT01827358
Title: Safety and Efficacy of Intranasal and Topical Mupirocin in Eradicating Colonization With Staphylococcus Aureus (SA) in Critically Ill Infants - a Phase 2, Multi-Center, Open Label, Randomized Trial
Brief Title: Safety and Efficacy of Mupirocin in Eradicating Colonization With S. Aureus in Critically Ill Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Prevention
Other Study IDs: 09-0065
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2016-04-13

CONDITIONS: Staphylococcal Infection
Keywords: antibacterial agent; children; colonisation; critically ill; infants; mupirocin; prevention; Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections; Critical Illness | interventions — Mupirocin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Subjects receive a 5-day course of mupirocin calcium ointment 2 % 20 mg intranasally applied every 8 hours and a topical skin application (umbilical and perianal area) of mupirocin calcium cream 2% 20 mg applied every 8 hours for a total of 15 doses
  Interventions: Drug: Mupirocin calcium
- Group 2 (No Intervention): No treatment

INTERVENTIONS:
Drug: Mupirocin calcium — Mupirocin calcium cream 2% applied topically to umbilicus and perianal area every 8 hours for 5 days, for a total of 15 applications
  Arms: Group 1
Drug: Mupirocin calcium — Mupirocin calcium ointment 2% will be applied intranasally every 8 hours for 5 days, for a total of 15 applications
  Arms: Group 1

SUMMARY:
The objective of this trial is 1) to evaluate the safety and clinical acceptability of a 5-day course of mupirocin applied every 8 hours (± 2 hours) to the nares, umbilical and perianal areas of infants residing in the ICU. 2) to examine the efficacy of mupirocin in eradicating SA colonization of infants in the ICU, defined as the absence of SA in cultures of the nares, umbilical, and perianal areas on day 8 (± 2) (primary decolonization) 3) to examine the efficacy of mupirocin in achieving persistent eradication of SA colonization among infants residing in the ICU,defined as the absence of SA in cultures of the nares, umbilical, and perianal areas. Duration is 36 months. Enrolled infants will continue to receive medical care as they otherwise would if they were not enrolled in the trial. The study will be powered with a primary endpoint with 126 participants. Enrollment may continue to 500 participants to power secondary and exploratory endpoints and assist design subsequent studies.

DETAILED DESCRIPTION:
This is a Phase 2, open label, multi-center, randomized trial to determine the safety and efficacy of mupirocin in eradicating colonization with Staphylococcus aureus (SA) and preventing the occurrence of invasive and other clinically significant SA infections among critically ill infants in the ICU. Infants hospitalized in an ICU at any one of the 6 participating centers with a positive nasal culture for SA will be eligible to enroll. Infants will be stratified by birth gestational age (< 28 weeks and <8 weeks of post-natal life or > /= 28 weeks / < 28 weeks and > /=8 weeks of post-natal life) and colonizing strain methicillin-resistant Staphylococcus aureus (MRSA) or methicillin-sensitive Staphylococcus aureus (MSSA) and then randomized 1:1 to receive a 5 day course of mupirocin applied to the nares, umbilicus and perianal (NUP) areas every 8 hours (± 2 hours) vs. no treatment. (Stratification by birth gestational age is performed to minimize bias that could result from a higher risk for developing infection due to prematurity or prolonged length of stay due to prematurity.) The primary objectives of this study are to 1) evaluate the safety and clinical acceptability of a 5-day course of mupirocin applied every 8 hours (± 2 hours) to the nares, umbilical and perianal areas of infants residing in the ICU 2) to examine the efficacy of mupirocin in eradicating SA colonization of infants in the ICU, defined as the absence of SA in cultures of the nares, umbilical, and perianal areas on day 8 (± 2) (primary decolonization) 3) to examine the efficacy of mupirocin in achieving persistent eradication of SA colonization among infants residing in the ICU, defined as the absence of SA in cultures of the nares, umbilical, and perianal areas on days 8 (±2) and 22 (±2) (persistent decolonization). The secondary objectives of this study are to 1) To examine the efficacy of mupirocin in preventing clinical SA infection during days 1-22 or until discharge, whichever occurs first, among SA colonized infants who are residing in the ICU 2) To compare time until SA decolonization between the mupirocin and placebo groups: Time from Day 1 until the first NUP collection with no SA is detected in the nares, umbilical, and perianal areas 3) To examine whether mupirocin affects the frequency of non-SA clinical infections by comparing the frequency of these infections in the treatment and control groups during the 85 day observation period 4) To examine whether mupirocin affects the frequency of severe (stage II-III) necrotizing enterocolitis by comparing the frequency of occurrence in the treatment and control groups during the 85 day observation period.

Each participant will be enrolled for up to 12 weeks (Day 85) or until the time of discharge from the hospital, death or withdrawal from further participation, whichever occurs first. It is anticipated that it will take at least 2 years to enroll all participants. Study duration is 36 months. Enrolled infants will continue to receive medical care as they otherwise would if they were not enrolled in the trial. The study will be powered toward the primary endpoint with 126 participants. Enrollment may continue up to a maximum of 500 participants to inform the secondary and exploratory endpoints and to help design any subsequent study.

ELIGIBILITY:
Inclusion Criteria:

1. Currently admitted to a NICU or ICU at a participating site 2. Chronological age less than 24 months 3. Evidence of colonization with SA (MRSA or MSSA) based on a positive nasal surveillance culture. Randomization must occur within 7 days (168 hours) of when the site's laboratory reports the first SA positive nasal surveillance swab 4. The attending neonatologist/ intensivist anticipates that the infant will remain in the ICU for a minimum of 14 days after enrollment 5. Parent or legal guardian agrees that the infant will not participate in a research trial involving the administration of an investigational drug for 14 days following enrollment

Exclusion Criteria:

1. Receipt of an investigational drug as part of a research trial within the past 14 days 2. Previously enrolled and participated in this trial 3. Has an active or previous SA infection 4. Currently receiving topical or intranasal mupirocin 5. Has a rash in an area to which mupirocin will be directly applied 6. Has any of the following congenital abnormalities: --A congenital skin disorder (i.e. - epidermolysis bullosa, icthyosis) --An opened neural tube defect --Confirmed or suspected choanal atresia --Any of the following abdominal wall defects: wound dehiscence, gastroschisis, open abdominal wound (small abdominal wall defects such as ostomy sites or peritoneal drain sites are not exclusionary) 7. Is nasally intubated 8. Known hypersensitivity to the trial product or its constituents 9. Known or suspected immune deficiency. Infants born to HIV-seropositive mothers with the following risk factors for intrapartum transmission will not be eligible to participate: --Mother's most recent viral load within the past 3 months was > 1,000 copies/ml or --Mother's viral load is not known or has has not been measured in the past 3 months. 10. Any other condition(s) that in the opinion of the investigator would jeopardize the safety or rights of a participant or would render the participant unable to comply with the protocol

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2014-04-30; Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Emory University Hospital Midtown - Neonatal Intensive Care Unit, Atlanta, Georgia
  - University of Maryland Medical Center - Children's Hospital - Neonatal Intensive Care Unit, Baltimore, Maryland
  - Children's Mercy Hospital and Clinics - Infectious Diseases, Kansas City, Missouri
  - Saint Louis University School of Medicine - Cardinal Glennon Children's Medical Center - NICU, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee

REFERENCES:
- [Derived] Kotloff KL, Shirley DT, Creech CB, Frey SE, Harrison CJ, Staat M, Anderson EJ, Dulkerian S, Thomsen IP, Al-Hosni M, Pahud BA, Bernstein DI, Yi J, Petrikin JE, Haberman B, Stephens K, Stephens I, Oler RE Jr, Conrad TM. Mupirocin for Staphylococcus aureus Decolonization of Infants in Neonatal Intensive Care Units. Pediatrics. 2019 Jan;143(1):e20181565. doi: 10.1542/peds.2018-1565. PMID 30587533

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants less than 24 months of age were recruited from among those admitted to the NICU or ICU at one of the participating centers found to have a surveillance nasal swab culture positive for SA. Recruitment was performed sequentially as infants became eligible without regards for race, ethnicity, gestational age or gender.
Pre-assignment Details: Infants were screened for nasal SA colonization (MRSA or MSSA) and only those who were colonized (not infected) were offered enrollment.
Groups:
- Mupirocin (Treatment): Participants received a 5-day course of mupirocin calcium ointment 2 % 20 mg intranasally applied every 8 hours and a topical skin application (umbilical and perianal area) of mupirocin calcium cream 2% 20 mg applied every 8 hours for a total of 15 doses
- No Mupirocin (Control): Participants received no treatment or placebo
Period: Overall Study
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Started | 80 | 75
Completed | 45 | 44
Not Completed | 35 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control) | Total
Number analyzed (Participants) | 80 | 75 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 80 | 75 | 155
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 4.6 (3.6) | 4.8 (4.4) | 4.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 33 | 68
  Male | 45 | 42 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 76 | 66 | 142
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 25 | 47
  White | 50 | 41 | 91
  More than one race | 6 | 7 | 13
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 80 | 75 | 155

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events (AEs) During Days 1-7
Description: Participants were evaluated for solicited adverse events while in the NICU/ICU on days 1-7. Participants were counted if they experienced the symptom at any severity during the reporting period. Although participants received only 5 days of mupirocin, solicited events were collected through day 7.
Time Frame: Days 1 through 7
Population: The analysis population was comprised of all infants, categorized according to treatment group. The number of infants is different from the overall study participant counts as 2 participants randomized to the mupirocin group received no mupirocin. For the purpose of safety analysis, these were included in the control (no mupirocin) group.
Measure: Number; unit: participants
Groups:
- No Mupirocin (Control): Participants received no treatment and no placebo.
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 78 | 77
participants
  Fever | 2 | 1
  Rash | 17 | 4
  Swelling of nasal mucosa | 1 | 0
  Epistaxis | 0 | 0
  Diarrhea | 9 | 7
  Apnea/ bradycardia/ desaturation events | 43 | 45
  Apnea within 3-5 minutes of mupirocin application | 8 | NA — Participants in the No Mupirocin (Control) group did not receive mupirocin
  Pain within 3-5 minutes of mupirocin application | 15 | NA — Participants in the No Mupirocin (Control) group did not receive mupirocin
  Any Symptom | 60 | 65

2. Primary Outcome: Number of Participants With Moderate and Severe Unsolicited Adverse Events; During Days 1-7
Description: Participants were evaluated for moderate and severe unsolicited adverse events (that were not otherwise considered pre-defined trial endpoints) while in the NICU/ICU on days 1-7. Although participants received 5 days of mupirocin, unsolicited events were collected until day 7. Moderate events were defined as those that may cause some interference with functioning and daily activities. Severe events were defined as those that interrupt the participant's usual daily activities and may require systemic drug therapy or other treatment. Severe events were usually incapacitating.
Time Frame: Days 1 through 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 78 | 77
participants
  Cardiac failure | 1 [0 to 7] | 0 [0 to 5]
  Heart disease congenital | 1 [0 to 7] | 0 [0 to 5]
  Incarcerated inguinal hernia | 1 [0 to 7] | 0 [0 to 5]
  Necrotising colitis | 0 [0 to 5] | 1 [0 to 7]
  Candida infection | 1 [0 to 7] | 0 [0 to 5]
  Pneumonia | 1 [0 to 7] | 0 [0 to 5]
  Rhinovirus infection | 0 [0 to 5] | 1 [0 to 7]

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) During Days 1-7
Description: Participants were evaluated for Serious Adverse Events (SAEs) while in the NICU/ICU on days 1-7. Although participants received only 5 days of mupirocin, SAEs were collected through day 7. An adverse event or suspected adverse reaction was considered serious if, in the view of either the investigator or sponsor, it resulted in any of the following outcomes: death; a life-threatening adverse event (an event that places the participant at immediate risk of death; it doesn't include an adverse event, had it occurred in a more severe form, might have caused death); inpatient hospitalization or prolongation of existing hospitalization; a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; or any other event that when based upon appropriate medical judgement may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Days 1 through 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 78 | 77
Participants
  Staphylococcal bacteremia | 1 | 0
  Heart disease congenital | 1 | 0
  Incarcerated inguinal hernia | 1 | 0
  Infantile apnoea | 1 | 0

4. Primary Outcome: Primary Decolonization Efficacy- Number of Participants in the Treatment and Control Groups Who Have no Detectable S. Aureus (SA) on Direct Nasal, Umbilical, and Perianal (NUP) Cultures Obtained on Day 8.
Description: Colonization was defined as the presence of SA identified by NUP culture without signs of illness or infection. On day 8, participants were swabbed in each of three areas: nasal, umbilical, and perianal. These swabs were cultured by direct plating. If SA did not grow on any of these cultures the infant was considered to be decolonized. If SA grew on any one of these cultures the infant was considered to be colonized with SA.
Time Frame: Day 8
Population: The analysis population included all infants with a site-specific pre-randomization NUP culture that was positive for SA by direct culture and who either had a complete set of NUP cultures collected on Day 8 or else had discontinued NUP cultures prior to day 8 due to a clinical SA infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 66 | 64
Participants | 62 | 3
Statistical Analysis 1: Comparison: Mupirocin (Treatment); Test type: Other — For strong control of the family-wise error rate at the 0.05 confidence level, the Holm procedure (Holm 1979) is used. Under this procedure, the p-values from the two tests are sorted as p_((1)) (smaller p-value) and p_((2)) (larger p-value). If p_((1))=0.025 and p_((2))=0.05, then the null hypotheses for both tests are rejected. If p_((1))=0.025 and p_((2))>0.05, then only the null hypothesis associated with the smaller p-value is rejected. In any other case, neither null hypothesis is rejected; p < 0.001, Fisher Exact; Odds Ratio (OR) = 315.2, 97.5% CI 2-sided [49.6 to 2698.8]

5. Primary Outcome: Persistent Decolonization Efficacy- Number of Participants in the Treatment and Control Groups Who Have no Detectable S. Aureus (SA) on Direct Nasal, Umbilical, and Perianal (NUP) Cultures on Days 8 and 22.
Description: Participants were admitted into the study based on being colonized with SA. Participants who were decolonized both on day 8 and day 22, as determined by NUP cultures were considered to have persistent decolonization. Colonization was defined as the presence of SA identified by NUP culture without signs of illness or infection. NUP swabs were collected on day 8 and on day 22 and cultured by direct plating. If the cultures were negative for SA at both day 8 and day 22 the participant was considered to have persistent decolonization. Colonization with SA was a prerequisite for enrollment, because of this there was no baseline measure.
Time Frame: Day 8 and Day 22
Population: The analysis population included all infants with a site-specific pre-randomization NUP culture that was positive for SA by direct culture and who had either had complete sets of NUP cultures collected on day 8 and day 22 or else had discontinued NUP cultures prior to day 22 due to a clinical SA infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 46 | 48
Participants | 21 | 1
Statistical Analysis 1: Comparison: Mupirocin (Treatment); Test type: Other — [test comment as in outcome 4, analysis 1]; p < 0.001, Fisher Exact; Odds Ratio (OR) = 39.5, 95% CI 2-sided [5.5 to 1666.3]

6. Secondary Outcome: Relative Risk of Occurrence of Non-SA Clinical Infection in the Treatment Compared to Control Group in the Intent To Treat Cohort
Description: Relative risk of occurrence of non-SA clinical infection in the treatment compared to the control group using the intent to treat (ITT) cohort for analysis. The time periods in the table correspond to the study days having scheduled collection of nasal, umbilical, and perianal (NUP) cultures. At risk participants were eligible for the non-SA clinical infection to occur at the start of the interval, were still on study and had not yet had a non-SA clinical infection but were still being watched for the event. Non-SA clinical infection was the development of a non-SA clinical infection due to an identifiable organism as evidenced by culture of an organism other than SA from a normally sterile body site or an infant who met the clinical diagnosis of localized infection as defined in the protocol. Censored participants were at risk for some of the interval, did not have a non-SA clinical infection but were removed from eligibility for the event at some point after the interval started.
Time Frame: Day 1 through 85
Population: The ITT cohort included all randomized infants. The analyses on the ITT cohort were performed per randomized treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 80 | 75
Participants
  Day 1-8 at risk | 78 | 73
  Day 1-8 with clinical non-SA infection | 3 | 1
  Day 1-8 censored | 4 | 6
  Day 9-15 at risk | 71 | 66
  Day 9-15 with clinical non-SA infection | 0 | 0
  Day 9-15 censored | 11 | 12
  Day 16-22 at risk | 60 | 54
  Day 16-22 with clinical non-SA infection | 0 | 0
  Day 16-22 censored | 12 | 4
  Day 23-29 at risk | 48 | 50
  Day 23-29 with clinical non-SA infection | 0 | 3
  Day 23-29 censored | 4 | 14
  Day 30-36 at risk | 44 | 33
  Day 30-36 with clinical non-SA infection | 1 | 1
  Day 30-36 censored | 6 | 6
  Day 37-43 at risk | 37 | 26
  Day 37-43 with clinical non-SA infection | 1 | 0
  Day 37-43 censored | 4 | 7
  Day 44-50 at risk | 32 | 19
  Day 44-50 with clinical non-SA infection | 0 | 0
  Day 44-50 censored | 9 | 6
  Day 51-57 at risk | 23 | 13
  Day 51-57 with clinical non-SA infection | 1 | 0
  Day 51-57 censored | 0 | 3
  Day 58-64 at risk | 22 | 10
  Day 58-64 with clinical non-SA infection | 0 | 0
  Day 58-64 censored | 5 | 5
  Day 65-71 at risk | 17 | 5
  Day 65-71 with clinical non-SA infection | 0 | 0
  Day 65-71 censored | 6 | 1
  Day 72-78 at risk | 11 | 4
  Day 72-78 with clinical non-SA infection | 0 | 0
  Day 72-78 censored | 3 | 0
  Day 79-85 at risk | 8 | 4
  Day 79-85 with clinical non-SA infection | 0 | 0
  Day 79-85 censored | 8 | 4
Statistical Analysis 1: Comparison: Mupirocin (Treatment); The association between mupirocin treatment and non-clinical SA Infection on or before Day 85 was assessed via a Cox Proportional Hazards Model. Onset time was defined as the first day of non-SA infection. Infants were right-censored at the time of discharge from the hospital or at Day 85, whichever came first; Test type: Other; p = 0.997, Cox proportional hazards model; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.30 to 3.28]

7. Secondary Outcome: Relative Risk of Occurrence of Non-SA Clinical Infection in the Treatment Compared to Control Group in the According to Protocol Cohort.
Description: Relative risk of occurrence of non-SA clinical infection in the treatment compared to control groups using the according to protocol (ATP) cohort. The time periods in the table correspond to the study days having scheduled collection of nasal, umbilical, and perianal (NUP) cultures. At risk participants were eligible for the non-SA clinical infection to occur at the start of the interval, were still on study and had not yet had a non-SA clinical infection but were still being watched for the event. Non-SA clinical infection was the development of a non-SA clinical infection due to an identifiable organism as evidenced by culture of an organism other than SA from a normally sterile body site or an infant who met the clinical diagnosis of localized infection as defined in the protocol. Censored participants were at risk for some of the interval, did not have a non-SA clinical infection but were removed from eligibility for the event at some point after the interval started.
Time Frame: Day 1 through 85
Population: The ATP cohort includes all infants with a site-specific pre-randomization NUP culture that is positive for SA by direct culture, those in the mupirocin treatment group must have received a minimum of 10 complete mupirocin treatments, including at least one dose to all three NUP sites per day for five consecutive days during the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 67 | 66
Participants
  Day 1-8 at risk | 67 | 66
  Day 1-8 with clinical non-SA infection | 3 | 1
  Day 1-8 censored | 3 | 4
  Day 9-15 at Risk | 61 | 61
  Day 9-15 with clinical non-SA infection | 0 | 0
  Day 9-15 censored | 9 | 11
  Day 16-22 at risk | 52 | 50
  Day 16-22 with non-SA infection | 0 | 0
  Day 16-22 censored | 11 | 4
  Day 23-29 at risk | 41 | 46
  Day 23-29 with clinical non-SA infection | 0 | 3
  Day 23-29 censored | 4 | 13
  Day 30-36 at risk | 37 | 30
  Day 30-36 with clinical non-SA infection | 1 | 0
  Day 30-36 censored | 4 | 6
  Day 37-43 at risk | 32 | 24
  Day 37-43 with clinical non-SA infection | 1 | 0
  Day 37-43 censored | 4 | 7
  Day 44-50 at risk | 27 | 17
  Day 44-50 with clinical non-SA infection | 0 | 0
  Day 44-50 censored | 8 | 6
  Day 51-57 at risk | 19 | 11
  Day 51-57 with clinical non-SA infection | 1 | 0
  Day 51-57 censored | 0 | 2
  Day 58-64 at risk | 18 | 9
  Day 58-64 with clinical non-SA infection | 0 | 0
  Day 58-64 censored | 4 | 4
  Day 65-71 at risk | 14 | 5
  Day 65-71 with clinical non-SA infection | 0 | 0
  Day 65-71 censored | 5 | 1
  Day 72-78 at risk | 9 | 4
  Day 72-78 with clinical non-SA infection | 0 | 0
  Day 72-78 censored | 3 | 0
  Day 79-85 at risk | 6 | 4
  Day 79-85 with clinical non-SA infection | 0 | 0
  Day 79-85 censored | 6 | 4
Statistical Analysis 1: Comparison: Mupirocin (Treatment); [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.656, Cox proportional hazards model; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.37 to 4.76]

8. Secondary Outcome: Median Time to Occurrence of Severe (Stage II-III) Necrotizing Enterocolitis (NEC) in the Treatment Compared to Control Group.
Description: Median time to occurrence of severe (stage II-III) NEC in the treatment compared to control group as estimated using Kaplan-Meier estimates of the survival curves.
Time Frame: Day 1 through 85
Population: There were no events of necrotizing enterocolitis during the study, analysis could not be performed.
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Protective Efficacy of Clinical S. Aureus (SA) Infection in the Treatment Compared to the Control Group During Days 1-22 or Until Discharge, Whichever Occurs First, Using the Intent to Treat Cohort.
Description: Protective efficacy of clinical SA infection in the treatment compared to the control group during days 1-22 or until discharge, whichever occurs first using the intent to treat (ITT) cohort. The time periods in the table correspond to the study days having scheduled collection of nasal, umbilical, and perianal (NUP) cultures. At risk participants were eligible for the SA clinical infection to occur at the start of the interval, were still on study and had not yet had a SA clinical infection but were still being watched for the event. SA clinical infection was the development of a SA clinical infection due to an identifiable organism as evidenced by culture of an organism from a normally sterile body site or an infant who met the clinical diagnosis of localized infection as defined in the protocol. Censored participants were at risk for some of the interval, did not have a SA clinical infection but were removed from eligibility for the event at some point after the interval started.
Time Frame: Day 1 through 22
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 80 | 75
Participants
  Day 1-8 at risk | 78 | 73
  Day 1-8 with clinical SA infection | 0 | 2
  Day 1-8 censored | 5 | 6
  Day 9-15 at risk | 73 | 65
  Day 9-15 with clinical SA infection | 1 | 1
  Day 9-15 censored | 11 | 12
  Day 16-22 at risk | 61 | 52
  Day 16-22 with clinical SA infection | 0 | 1
  Day 16-22 censored | 61 | 51
Statistical Analysis 1: Comparison: Mupirocin (Treatment); The time to clinical infection with SA on or prior to Day 22 was analyzed using Kaplan-Meier estimates of the survival curve and Cox proportional hazards models (with treatment as the only independent variable). Infants were censored at Day 22 or completion or early termination from the study. Estimates of the hazard ratio (values less than one indicating a treatment benefit) with Wald 95% confidence intervals and accompanying p-values were calculated; Test type: Other; p = 0.182, Cox proportional hazards models; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.03 to 2.01]

10. Secondary Outcome: Protective Efficacy of Clinical SA Infection in the Treatment Compared to the Control Group During Days 1-22 or Until Discharge, Whichever Occurs First, Using the According to Protocol (ATP) Cohort.
Description: Protective efficacy of clinical SA infection in the treatment compared to the control group during days 1-22 or until discharge, whichever occurs first using the ATP cohort. The time periods in the table correspond to the study days having scheduled collection of nasal, umbilical, and perianal (NUP) cultures. At risk participants were eligible for the SA clinical infection to occur at the start of the interval, were still on study and had not yet had a SA clinical infection but were still being watched for the event. SA clinical infection was the development of a SA clinical infection due to an identifiable organism as evidenced by culture of an organism from a normally sterile body site or an infant who met the clinical diagnosis of localized infection as defined in the protocol. Censored participants were at risk for some of the interval, did not have a SA clinical infection but were removed from eligibility for the event at some point after the interval started.
Time Frame: Day 1 through 22
Population: The ATP cohort includes all infants that have met all requirements of the mITT cohort, with the further requirements that infants in the mupirocin treatment group must have received a minimum of 10 complete mupirocin treatments, including at least one dose to all three NUP sites per day for five consecutive days during the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 67 | 66
Participants
  Day 1-8 at risk | 67 | 66
  Day 1-8 with clinical SA infection | 0 | 2
  Day 1-8 censored | 4 | 4
  Day 9-15 at risk | 63 | 60
  Day 9-15 with clinical SA infection | 1 | 1
  Day 9-15 censored | 9 | 11
  Day 16-22 at risk | 53 | 48
  Day 16-22 with clinical SA infection | 0 | 1
  Day 16-22 censored | 53 | 47
Statistical Analysis 1: Comparison: Mupirocin (Treatment); [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.198, Cox proportional hazards model; Hazard Ratio (HR) = 0.24, 95% CI 2-sided [0.03 to 2.12]

11. Secondary Outcome: Median Time to Occurrence of Non-S. Aureus (SA) Clinical Infection in the Treatment Compared to Control Group
Description: Median time to occurrence of non-SA clinical infection in the treatment compared to control group as estimated using Kaplan-Meier estimates of the survival curves.
Time Frame: Day 1 through 85
Population: Clinical infection besides SA infection on or prior to Day 85 was not observed frequently enough to allow estimation of the median time to infection using non-parametric methods.
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Relative Risk of Severe (Stage II-III) Necrotizing Enterocolitis (NEC) in the Treatment Compared to Control Group
Description: The association between mupirocin treatment and severe (stage II-III) NEC on or before Day 85 was to be assessed via Cox Proportional Hazards Model.
Time Frame: Day 1 through 85
Population: There were no events of necrotizing enterocolitis during the study, analysis could not be performed.
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Time Until Decolonization: Count of Participants From Day 1 Until the First NUP Collection With no S. Aureus (SA) Detected in the Nares, Umbilical, and Perianal Areas Using the Modified Intent to Treat Day 8 Cohort (mITT-8).
Description: Time until decolonization: Count of participants from Day 1 until the first NUP collection with no SA is detected in the nares, umbilical, and perianal areas using the modified intent to treat (mITT-8) cohort. The time periods in the table correspond to the study days having collection of nasal, umbilical, and perianal (NUP) cultures. At risk participants were eligible for the SA decolonization to occur at the start of the interval, were still on study and had not yet had SA decolonization but were still being watched for the event. SA decolonization was the absence of SA detected from the NUP cultures through direct plating. Censored participants were at risk for some of the interval, did not have SA decolonization but were removed from eligibility for the event at some point after the interval started.
Time Frame: Day 1 through 85
Population: The mITT cohort includes all infants with a site-specific pre-randomization NUP culture that was positive for SA by direct culture. The mITT-8 cohort includes all mITT infants who either had a complete set of NUP cultures collected on day 8 or else had discontinuation of NUP cultures prior to Day 8 due to a clinical SA infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 66 | 64
Participants
  Day 1-8 at risk | 66 | 64
  Day 1-8 with decolonization | 59 | 3
  Day 1-8 censored | 1 | 14
  Day 9-15 at risk | 6 | 47
  Day 9-15 with decolonization | 3 | 0
  Day 9-15 censored | 0 | 4
  Day 16-22 at risk | 3 | 43
  Day 16-22 with decolonization | 0 | 0
  Day 16-22 censored | 3 | 43

14. Secondary Outcome: Time Until Decolonization: Count of Participants From Day 1 Until the First NUP Collection With no SA is Detected in the Nares, Umbilical, and Perianal Areas Using the According to Protocol Day 8 (ATP-8) Cohort.
Description: Time until decolonization: Count of participants from Day 1 until the first NUP collection with no SA is detected in the nares, umbilical, and perianal areas using the according to protocol day 8 (ATP-8) cohort. The time periods in the table correspond to the study days having scheduled collection of nasal, umbilical, and perianal (NUP) cultures. At risk participants were eligible for the SA decolonization to occur at the start of the interval, were still on study and had not yet had SA decolonization but were still being watched for the event. SA decolonization was the absence of SA detected from the NUP cultures through direct plating. Censored participants were at risk for some of the interval, did not have SA decolonization but were removed from eligibility for the event at some point after the interval started.
Time Frame: Day 1 through 85
Population: The ATP-8 cohort includes all ATP infants who had a set of NUP cultures collected on Day 8 (± 2).
Measure: Count of Participants; unit: Participants
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Number analyzed (Participants) | 64 | 63
Participants
  Day 1-8 at risk | 64 | 63
  Day 1-8 with decolonization | 57 | 2
  Day 1-8 censored | 1 | 14
  Day 9-15 at risk | 6 | 47
  Day 9-15 with decolonization | 3 | 0
  Day 9-15 censored | 0 | 4
  Day 16-22 at risk | 3 | 43
  Day 16-22 with decolonization | 0 | 0
  Day 16-22 censored | 3 | 43

ADVERSE EVENTS:
Time Frame: Adverse events were collected on days 1-7.
Description: For days 1-7, study staff were responsible for identifying solicited adverse events (AEs), unsolicited moderate and severe AEs and serious adverse events (SAEs) on a daily basis. Solicited adverse events of apnea within 3-5 minutes of mupirocin application and pain within 3-5 minutes of mupirocin application, were not applicable to the control group since they did not receive mupirocin.
Groups:
- Mupirocin (Treatment): Participants receive a 5-day course of mupirocin calcium ointment 2 % 20 mg intranasally applied every 8 hours and a topical skin application (umbilical and perianal area) of mupirocin calcium cream 2% 20 mg applied every 8 hours for a total of 15 doses
Arm/Group | Mupirocin (Treatment) | No Mupirocin (Control)
Serious Adverse Events (participants affected / at risk) | 3/80 | 0/75
Other Adverse Events (participants affected / at risk) | 60/78 | 50/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mupirocin (Treatment) (N=80) | No Mupirocin (Control) (N=75)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Mupirocin (Treatment) (N=78) | No Mupirocin (Control) (N=77)
Rash (Skin and subcutaneous tissue disorders) | 17 (52) | 4 (12)
Diarrhoea (Gastrointestinal disorders) | 9 (18) | 7 (14)
Apnea (Respiratory, thoracic and mediastinal disorders) | 43 (128) | 45 (129)
Administration related reaction (Injury, poisoning and procedural complications) | 8 (9) | 0/0 (0)
Application site pain (General disorders) | 15 (18) | 0/0 (0) — Administration site conditions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less